CLINICAL TRIAL: NCT03959241
Title: A Randomized, Multicenter, Phase III Trial of Tacrolimus/Methotrexate Versus Post-Transplant Cyclophosphamide/Tacrolimus/Mycophenolate Mofetil in Non-Myeloablative/Reduced Intensity Conditioning Allogeneic Peripheral Blood Stem Cell Transplantation (BMT CTN 1703; Progress III); Companion Study: Microbiome and Immune Reconstitution in Cellular Therapies and Hematopoietic Stem Cell Transplantation (BMT CTN 1801; Mi-Immune)
Brief Title: TAC/MTX vs. TAC/MMF/PTCY for Prevention of Graft-versus-Host Disease and Microbiome and Immune Reconstitution Study (BMT CTN 1703/1801)
Acronym: 1703/1801
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BMT CTN 1703/1801; 2U10HL069294-11 (NIH)
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Results first posted 2024-01-12 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Acute Leukemia; Chronic Myelogenous Leukemia (CML); Myelodysplasia; Lymphoma
Keywords: Acute Leukemia; Chronic Myelogenous Leukemia (CML); Myelodysplasia (MDS); Lymphoma; GVHD prophylaxis; Acute GVHD
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Anemia, Refractory, with Excess of Blasts; Lymphoma | interventions — Tacrolimus; Methotrexate; Mycophenolic Acid; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Patients will be randomized at a ratio of 1:1 between the treatment arms using permuted blocks of random sizes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus/Methotrexate (Active Comparator): Mobilized Peripheral Blood Stem Cell graft with Tacrolimus/Methotrexate
  Interventions: Procedure: Mobilized Peripheral Blood Stem Cell graft with Tacrolimus/Methotrexate; Drug: Tacrolimus; Drug: Methotrexate
- Tacrolimus/MMF/PTCY (Experimental): Mobilized Peripheral Blood Stem Cell graft with Tacrolimus/Mycophenolate Mofetil/Post-Transplant Cyclophosphamide
  Interventions: Procedure: Mobilized Peripheral Blood Stem Cell graft with Tacrolimus/Mycophenolate Mofetil/Post-Transplant Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: Cyclophosphamide

INTERVENTIONS:
Procedure: Mobilized Peripheral Blood Stem Cell graft with Tacrolimus/Methotrexate — Mobilized PBSC grafts will be administered on Day 0 to all patients according to individual institutional guidelines after appropriate processing and quantification has been performed by the local laboratory. Stem cells are administered through an indwelling central venous catheter. If infusion occurs over two days, Day 0 is the first day the infusion is initiated.
  Other Names: HSCT
  Arms: Tacrolimus/Methotrexate
Drug: Tacrolimus — Tacrolimus will be given per institutional practices, orally at a dose of 0.05-0.06 mg/kg/day or intravenously at a dose of 0.02-0.03 mg/kg/day starting on Day -3. The dose of tacrolimus may be rounded to the nearest 0.5 mg for oral formulations. Subsequent dosing will be based on blood levels per institutional guidelines with a suggested range of 5-15. If patients are on medications which alter the metabolism of tacrolimus (e.g.concurrent CYP3A4 inhibitors), the initial starting dose and subsequent doses should be altered as per institutional practices. Tacrolimus taper can be initiated at a minimum of 90 days post HCT if there is no evidence of active GVHD. The rate of tapering will be done according institutional practices and patients should be off tacrolimus by Day 180 post HCT if there is no evidence of active GVHD.
  Other Names: Prograf®; FK506
  Arms: Tacrolimus/Methotrexate
Drug: Methotrexate — Methotrexate will be administered at the doses of 15 mg/m2 IV bolus on Day +1, and 10 mg/m2 IV bolus on Days +3, +6 and +11 after hematopoietic stem cell infusion. Methotrexate should be dose reduced, given with leucovorin rescue, or held for complications such as severe mucositis per institutional guidelines.
  Other Names: MTX
  Arms: Tacrolimus/Methotrexate
Procedure: Mobilized Peripheral Blood Stem Cell graft with Tacrolimus/Mycophenolate Mofetil/Post-Transplant Cyclophosphamide — Mobilized PBSC grafts will be administered on Day 0 to all patients according to individual institutional guidelines after appropriate processing and quantification has been performed by the local laboratory. Stem cells are administered through an indwelling central venous catheter. If infusion occurs over two days, Day 0 is the first day the infusion is initiated.
  Other Names: HSCT
  Arms: Tacrolimus/MMF/PTCY
Drug: Tacrolimus — Tacrolimus will be given per institutional practices, orally at a dose of 0.05-0.06 mg/kg/day or intravenously at a dose of 0.02-0.03 mg/kg/day starting Day +5. Starting tacrolimus dose can be modified to account for possible drug interactions (e.g. concurrent CYP3A4 inhibitor use) according to institutional guides. Serum levels of tacrolimus will be measured at Day +7 and then should be checked weekly thereafter, and the dose adjusted accordingly to maintain a suggested level of 5-15 ng/mL. Tacrolimus taper can be initiated at a minimum of 90 days post HCT if there is no evidence of active GVHD. The rate of tapering will be done according to institutional practices but patients should be off tacrolimus by Day 180 post HCT if there is no evidence of active GVHD
  Other Names: Prograf®; FK506
  Arms: Tacrolimus/MMF/PTCY
Drug: Mycophenolate Mofetil — MMF will be given at a dose of 15 mg/kg/dose ter in die (TID) (based upon actual body weight) with the maximum total daily dose not to exceed 3 grams (1g TID, IV or PO). MMF prophylaxis will start Day +5 and discontinue after the last dose on Day +35, or may be continued if active GVHD is present.
  Other Names: CellCept®; MMF
  Arms: Tacrolimus/MMF/PTCY
Drug: Cyclophosphamide — Cyclophosphamide [50 mg/kg ideal body weight (IBW); if actual body weight (ABW) < IBW, use ABW] will be given on Day +3 (between 60 and 72 hours after the start of the PBSC infusion) and on Day +4 post-transplant (approximately 24 hours after Day +3 cyclophosphamide). Cyclophosphamide will be given as an IV infusion over 1-2 hours (depending on volume).
  Other Names: Cytoxan®
  Arms: Tacrolimus/MMF/PTCY

SUMMARY:
1703: The study is designed as a randomized, phase III, multicenter trial comparing two acute graft-versus-host disease (aGVHD) prophylaxis regimens: tacrolimus/methotrexate (Tac/MTX) versus post-transplant cyclophosphamide/tacrolimus/mycophenolate mofetil (PTCy/Tac/MMF) in the setting of reduced intensity conditioning (RIC) allogeneic peripheral blood stem cell (PBSC) transplantation.

1801: The goal of this protocol is to test the primary hypothesis that the engraftment stool microbiome diversity predicts one-year non-relapse mortality in patients undergoing reduced intensity allogeneic HCT.

DETAILED DESCRIPTION:
1703: Graft-versus-Host Disease (GVHD) is a complication that affects many hematopoietic stem cell transplant (HSCT) patients; it occurs when the new cells from a transplant attack the recipient's body. The current standard GVHD prophylaxis regimen for patients with hematologic malignancies undergoing HSCT involves a combination of immunosuppressive agents given for the first 6 months after transplant.

The standard strategy of Tacrolimus/Methotrexate will be used as a control arm in comparison to one other treatment plan utilizing Tacrolimus/Mycophenolate Mofetil/Post-Transplant Cyclophosphamide. Study participants will receive an infusion of mobilized peripheral blood stem cell grafts on both arms. Study participants will be randomized to one of these two treatment arms.

1801: A relationship between the intestinal microbiota and graft-versus-host disease (GVHD) has long been appreciated but is still not well understood. Mice transplanted in germ-free conditions or treated with gut-decontaminating antibiotics developed less severe GVHD. Clinical studies initially suggested a benefit from near-total bacterial decontamination, but later showed no clear benefit and this approach was discontinued in the early 1990s. Partial gut decontamination continues to be practiced at many centers. More recently, the advent of next-generation sequencing (NGS) has resulted in cheaper and easier characterization of complex microbial mixtures. This has led to a renewed interest in evaluating the relationship between the microbiota and human health and disease, including recipients of hematopoietic cell transplantation (HCT). Similarly, NGS has also contributed to significant advancements in the investigator's understanding of immune reconstitution in HCT patients and how this may impact clinica outcomes.

The goal of this protocol is to test the primary hypothesis that the engraftment stool microbiome diversity predicts one-year non-relapse mortality in patients undergoing reduced intensity allogeneic HCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18.0 years or older at the time of enrollment on Segment A
2. Patients with acute leukemia or chronic myelogenous leukemia with no circulating blasts and with less than 5% blasts in the bone marrow
3. Patients with myelodysplasia/chronic myelomonocytic leukemia with no circulating blasts and with less than 10% blasts in the bone marrow (higher blast percentage allowed in MDS due to lack of differences in outcomes with <5% vs. 5-10% blasts in this disease)
4. Patients with relapsed chronic lymphocytic leukemia/small lymphocytic lymphoma with chemosensitive disease at time of transplantation
5. Patients with lymphoma [follicular lymphoma, Hodgkin lymphoma, diffuse large B cell lymphoma, mantle cell lymphoma, peripheral T-cell lymphoma, angioimmunoblastic T-cell lymphoma and anaplastic large cell lymphoma] with chemosensitive disease at the time of transplantation
6. Planned reduced intensity conditioning regimen (see eligible regimens in Table 2.4a)
7. Patients must have a related or unrelated peripheral blood stem cell donor as follows:

   1. Sibling donor must be a 6/6 match for Human Leukocyte Antigen-A (HLA)-A and -B at intermediate (or higher) resolution, and -DRB1 at high resolution using DNA-based typing, and must be willing to donate peripheral blood stem cells and meet institutional criteria for donation.
   2. Unrelated donor must be a 7/8 or 8/8 match at HLA-A, -B, -C and -DRB1 at high resolution using DNA-based typing. Unrelated donor must be willing to donate peripheral blood stem cells and meet National Marrow Donor Program (NMDP) criteria for donation.
8. Cardiac function: Left ventricular ejection fraction at least 45%
9. Estimated creatinine clearance acceptable per institutional guidelines
10. Pulmonary function: Diffusing capacity of lung for carbon monoxide (DLCO) corrected for hemoglobin at least 40% and forced expiratory volume at one second (FEV1) predicted at least 50%
11. Liver function acceptable per institutional guidelines
12. Karnofsky Performance Score at least 60%
13. Female patients (unless postmenopausal for at least 1 year before the screening visit, or surgically sterilized), agree to practice two (2) effective methods of contraception at the same time, or agree to completely abstain from heterosexual intercourse, from the time of signing the informed consent through 12 months post-transplant (see Section 2.6.4 for definition of postmenopausal)
14. Male patients (even if surgically sterilized), of partners of women of childbearing potential must agree to one of the following: practice effective barrier contraception (see Section 2.6.4 for list of barrier methods), or abstain from heterosexual intercourse from the time of signing the informed consent through 12 months post-transplant
15. Plans for the use of post-transplant maintenance therapy must be disclosed upon enrollment and must be used irrespective of the outcome of the randomization. Please note that THIS DOES NOT INCLUDE INVESTIGATIONAL AGENTS and maintenance therapy with investigational treatment requires approval by the study chairs.
16. Voluntary written consent obtained prior to the performance of any study-related procedure that is not a part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

1. Prior allogeneic transplant
2. Active central nervous system (CNS) involvement by malignant cells
3. Patients with secondary acute myeloid leukemia arising from myeloproliferative disease, including chronic myelomonocytic leukemia (CMML)
4. Patients with uncontrolled bacterial, viral or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment.
5. Presence of clinically significant fluid collection (ascites, pleural or pericardial effusion) that interferes with methotrexate clearance or makes methotrexate use contraindicated
6. Patients seropositive for human immunodeficiency virus (HIV) with detectable viral load. HIV+ patients with an undetectable viral load on antiviral therapy are eligible.
7. Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia.
8. Female patients who are pregnant (as per institutional practice) or lactating
9. Patients with a serious medical or psychiatric illness likely to interfere with participation in this clinical study
10. Patients with prior malignancies except resected non-melanoma skin cancer or treated cervical carcinoma in situ. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously must be reviewed and approved by the Protocol Officer or Chairs.
11. Planned use of antithymocyte globulin (ATG) or alemtuzumab in conditioning regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, MS, Study Director — Center for International Blood and Marrow Transplant Research
Locations (39):
- United States (39):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - University of California, San Francisco, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Blood & Marrow Transplant Program at Northside Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Loyola University, Maywood, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Indiana BMT - St. Francis Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute/Brigham & Women's, Boston, Massachusetts
  - Dana Farber Cancer Institute/Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State/Arthur G. James Cancer Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine/The Methodist Hospital, Houston, Texas
  - University of Texas, MD Anderson Cancer Research Center, Houston, Texas
  - Virginia Commonwealth University, MCV Hospital, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Background] Bolanos-Meade J, Hamadani M, Wu J, Al Malki MM, Martens MJ, Runaas L, Elmariah H, Rezvani AR, Gooptu M, Larkin KT, Shaffer BC, El Jurdi N, Loren AW, Solh M, Hall AC, Alousi AM, Jamy OH, Perales MA, Yao JM, Applegate K, Bhatt AS, Kean LS, Efebera YA, Reshef R, Clark W, DiFronzo NL, Leifer E, Horowitz MM, Jones RJ, Holtan SG; BMT CTN 1703 Investigators. Post-Transplantation Cyclophosphamide-Based Graft-versus-Host Disease Prophylaxis. N Engl J Med. 2023 Jun 22;388(25):2338-2348. doi: 10.1056/NEJMoa2215943. PMID 37342922
- [Derived] Abedin S, Martens MJ, Bolanos-Meade J, Al Malki MM, Lian Q, Runaas L, Elmariah H, Gooptu M, Larkin KT, Shaffer BC, Loren AW, Solh M, Alousi AM, Jamy OH, Perales MA, Rezvani A, Bhatt A, El Jurdi N, Yao JM, Applegate K, Kean LS, Efebera YA, Reshef R, Clark W, Leifer E, Saber W, Horowitz MM, Jones RJ, Holtan SG, Hamadani M. Impact of posttransplant cyclophosphamide-based GVHD prophylaxis in patients 70 years and older: an update from BMT CTN 1703. Blood Adv. 2025 Jul 22;9(14):3495-3501. doi: 10.1182/bloodadvances.2025015964. PMID 40305657
- [Derived] Holtan SG, Bolanos-Meade J, Al Malki MM, Wu J, Kitko CL, Reshef R, Rezvani AR, Shaffer BC, Solh MM, Yao JM, Runaas L, Elmariah H, Larkin KT, El Jurdi N, Gooptu M, Loren AW, Hall AC, Alousi AM, Jamy O, Clark W, Kean L, Bhatt AS, Perales MA, Applegate K, Efebera YA, Leifer E, Jones RJ, Horowitz MM, Mattila D, Saber W, Hamadani M, Martens MJ. Improved Patient-Reported Outcomes With Post-Transplant Cyclophosphamide: A Quality-of-Life Evaluation and 2-Year Outcomes of BMT CTN 1703. J Clin Oncol. 2025 Mar 10;43(8):912-918. doi: 10.1200/JCO.24.00921. Epub 2025 Jan 3. PMID 39752608
- See also: Blood and Marrow Transplant Clinical Trials Network Website — https://bmtctn.net//

RESULTS

PARTICIPANT FLOW:
Recruitment Details: BMT CTN 1703's enrollment was between June 2019 and June 2021 with 431 participants enrolled from 37 centers. The study opened to accrual on June 25, 2019 with 39 centers activated for enrollment. The study closed to accrual on June 18, 2021 and study completed on September 19, 2022.
  BMT CTN 1801 is a companion study to BMT CTN 1703. The accrual goal was 300 participants. Enrollment to BMT CTN 1801 is performed solely through co-enrollment of BMT CTN 1703 participants.
Pre-assignment Details: Enrolled participants were randomized in a 1:1 ratio to the two treatment arms. This is an open-label study and not blinded in treatment assignment. The randomized participants were intended to undergo transplant. For various reasons, a small portion of participants did not receive a transplant.
Groups:
- PTCY/Tacrolimus/MMF: Mobilized Peripheral Blood Stem Cell graft with Tacrolimus/Mycophenolate Mofetil/Post-Transplant Cyclophosphamide: Mobilized PBSC grafts will be administered on Day 0 to all patients. Stem cells are administered through an indwelling central venous catheter.
  Tacrolimus: Tacrolimus will be given per institutional practices, orally at a dose of 0.05-0.06 mg/kg/day or intravenously at a dose of 0.02-0.03 mg/kg/day starting Day +5. Serum levels of tacrolimus will be measured at Day +7 and then should be checked weekly thereafter, the dose adjusted accordingly to maintain a suggested level of 5-15 ng/mL. Tacrolimus taper can be initiated at 90 days post HCT if there is no evidence of active GVHD. The tapering rate will be based on institutional practices, patients should be off tacrolimus by Day 180 post HCT if there is no evidence of active GVHD.
  Mycophenolate Mofetil: MMF will be given at a dose of 15 mg/kg/dose ter in die (TID) with the maximum total daily dose not to exceed 3 grams (1g TID, IV or PO). MMF prophylaxis will start Day +5 and discontinue after the last dose on Day +35, or may be continued if active GVHD is present.
  Cyclophosphamide: Cyclophosphamide [50 mg/kg ideal body weight (IBW); if actual body weight (ABW) < IBW, use ABW] will be given on Day +3 (between 60 and 72 hours after the start of the PBSC infusion) and on Day +4 post-transplant (approximately 24 hours after Day +3 cyclophosphamide). Cyclophosphamide will be given as an IV infusion over 1-2 hours.
- Tacrolimus/Methotrexate: Mobilized Peripheral Blood Stem Cell graft with Tacrolimus/Methotrexate: Mobilized PBSC grafts will be administered on Day 0 to all patients according to individual institutional guidelines after appropriate processing and quantification has been performed by the local laboratory. Stem cells are administered through an indwelling central venous catheter. If infusion occurs over two days, Day 0 is the first day the infusion is initiated.
  Tacrolimus: Tacrolimus will be given per institutional practices, orally at a dose of 0.05-0.06 mg/kg/day or intravenously at a dose of 0.02-0.03 mg/kg/day starting on Day -3. Subsequent dosing will be based on blood levels per institutional guidelines with a suggested range of 5-15. If patients are on medications which alter the metabolism of tacrolimus, the initial starting dose and subsequent doses should be altered as per institutional practices. Tacrolimus taper can be initiated at a minimum of 90 days post HCT if there is no evidence of active GVHD. The rate of tapering will be done according institutional practices and patients should be off tacrolimus by Day 180 post HCT if there is no evidence of active GVHD.
  Methotrexate: Methotrexate will be administered at the doses of 15 mg/m2 IV bolus on Day +1, and 10 mg/m2 IV bolus on Days +3, +6 and +11 after hematopoietic stem cell infusion. Methotrexate should be dose reduced, given with leucovorin rescue, or held for complications such as severe mucositis per institutional guidelines.
Period: Overall Study
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Started | 214 | 217
Completed | 203 | 208
Not Completed | 11 | 9
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Lost to Follow-up | 1 | 0
Not completed — Move to Hospice Care | 1 | 0
Not completed — Screen Failure | 1 | 0
Not completed — Disease Relapse | 0 | 1
Not completed — Off Study | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate | Total
Number analyzed (Participants) | 214 | 217 | 431
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (8.5) | 64.5 (8.9) | 64.3 (8.7)
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 94 | 92 | 186
  65 years or older | 120 | 125 | 245
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 91 | 171
  Male | 134 | 126 | 260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 22 | 31
  Not Hispanic or Latino | 203 | 191 | 394
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 10 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 186 | 193 | 379
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 10 | 13 | 23
Karnofsky / Lansky Performance Score [Count of Participants; unit: Participants] — KPS describes patient-perceived global quality of life and functioning on a scale of 0-100.
  100: No evidence of disease; 90: Normal activity. Minor signs or symptoms of disease; 80: Normal activity with effort. Some signs or symptoms of disease; 70: Cares for self. Unable to continue normal activity; 60: Needs occasional assistance, but cares for most personal needs; 50: Needs considerable assistance and medical care; 40: Disabled. Needs special care and assistance; 30: Severely disabled. Hospital admission indicated; 20: Very sick. Active supportive therapy needed; 10: Moribund; 0: Dead
  Participants
    At least 90 | 106 | 108 | 214
    Less Than 90 | 108 | 109 | 217
Primary Disease [Count of Participants; unit: Participants]
  Acute lymphoblastic leukemia (ALL) | 12 | 27 | 39
  Acute myelogenous leukemia (AML) | 107 | 100 | 207
  Chronic myelogenous leukemia (CML) | 6 | 5 | 11
  Myelodysplastic syndrome (MDS) | 63 | 65 | 128
  Hodgkin lymphoma | 3 | 3 | 6
  Mantle cell lymphoma | 0 | 1 | 1
  Indolent NHL | 3 | 1 | 4
  T-cell NHL | 7 | 5 | 12
  Aggressive NHL | 9 | 7 | 16
  Burkitt lymphoma | 1 | 0 | 1
  Biphenotypic leukemia | 1 | 1 | 2
Time from Disease Diagnosis to Transplant [Mean (Standard Deviation); unit: months] | 12.3 (17.0) | 13.1 (21.5) | 12.7 (19.4)
Disease Risk Index [Count of Participants; unit: Participants] — The disease risk index (DRI) for allogeneic stem cell transplantation was assigned to participants based on the 2014 Refined Disease Risk Index. The refined DRI was validated using a multivariable regression model for overall survival. The classification table for identifying DRI group based on primary diagnosis, cytogenetics, and stage can be found in Appendix F of the study protocol. More severe DRI indicates higher risk.
  Participants
    Low | 19 | 21 | 40
    Intermediate | 125 | 125 | 250
    High / Very High | 70 | 71 | 141
Allogeneic Hematopoietic Cell Transplantation-Comorbidity Index (HCT-CI) total score [Count of Participants; unit: Participants] — HCT-CI identifies comorbidities relevant to transplant. Migraine, osteoporosis, osteoarthritis, hypertension, GI, mild pulmonary/renal, endocrine, and asthma are assigned a score of 0; Arrhythmia, cardiac, mild hepatic, diabetes, cerebrovascular, psychological, obesity, and infection a score 1; Rheumatologic, peptic ulcer, renal moderate/severe, and moderate pulmonary a score 2; Solid tumor, heart valve disease, severe pulmonary, and hepatic moderate/severe a score 3. The index score presented is the sum of all comorbidities present per patient. Scores >3 are combined in the 4+ category.
  Participants
    0 | 49 | 53 | 102
    1 | 31 | 34 | 65
    2 | 60 | 34 | 94
    3 | 24 | 33 | 57
    4+ | 40 | 55 | 95
    Missing/Unknown | 10 | 8 | 18
Donor Type and HLA Matching [Count of Participants; unit: Participants] — HLA Match Score includes genetic matching information at HLA-A, -B, and -DRB1 loci or HLA-A, -B, -C, and -DRB1 loci. Matching at all HLA-A, -B, and -DRB1 loci is designated as 6/6 HLA matching. A 4/6 HLA match includes mismatches at any two loci. Matching at all HLA-A, -B, -C, and -DRB1 loci is designated as 8/8 HLA matching. A 6/8 HLA match includes mismatches at any two loci.
  Participants
    Related donor 6/6 | 60 | 68 | 128
    Unrelated donor 7/8 | 7 | 8 | 15
    Unrelated donor 8/8 | 147 | 141 | 288
Donor/Recipient CMV Status [Count of Participants; unit: Participants]
  Pos/Pos | 61 | 71 | 132
  Pos/Neg | 20 | 32 | 52
  Neg/Pos | 67 | 40 | 107
  Neg/Neg | 59 | 70 | 129
  Missing/Unknown | 7 | 4 | 11
Donor/Recipient Sex Match [Count of Participants; unit: Participants]
  M-M | 85 | 75 | 160
  M-F | 41 | 54 | 95
  F-M | 47 | 49 | 96
  F-F | 36 | 35 | 71
  Missing/Unknown | 5 | 4 | 9
Donor/Recipient ABO Match [Count of Participants; unit: Participants] — Match is when donor blood type is the same as the recipient blood type; minor mismatch is donor O vs. recipient AB; major mismatch is donor AB vs. recipient O; the remainder are bi-directional mismatches.
  Participants
    Match | 122 | 111 | 233
    Minor Mismatch | 6 | 1 | 7
    Major Mismatch | 2 | 1 | 3
    Bidirectional Mismatch | 66 | 83 | 149
    Missing/Unknown | 18 | 21 | 39
Received reduced intensity conditioning regimen [Count of Participants; unit: Participants]
  Fludarabine/Busulfan | 56 | 61 | 117
  Fludarabine/Melphalan | 122 | 123 | 245
  Fludarabine/Cyclophosphamide | 5 | 1 | 6
  Fludarabine/TBI | 1 | 4 | 5
  Fludarabine/Cyclophosphamide/TBI | 24 | 24 | 48
  Missing/Unknown | 6 | 4 | 10
Planned Reduced Intensity Conditioning Regimen [Count of Participants; unit: Participants]
  Fludarabine/Busulfan | 58 | 61 | 119
  Fludarabine/Melphalan | 125 | 127 | 252
  Fludarabine/Cyclophosphamide | 6 | 1 | 7
  Fludarabine/TBI | 1 | 4 | 5
  Fludarabine/Cyclophosphamide/TBI | 24 | 24 | 48
Planned Post-Transplant Maintenance Therapy [Count of Participants; unit: Participants]
  No Planned Post-Transplant Maintenance Therapy | 159 | 170 | 329
  Tyrosine Kinase Inhibitor | 12 | 15 | 27
  FLT3 Inhibitor | 10 | 9 | 19
  Monoclonal Antibody | 1 | 0 | 1
  Clinical Trial | 1 | 1 | 2
  Other | 31 | 22 | 53

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With GVHD/Relapse or Progression-free Survival (GRFS) at One Year
Description: The primary endpoint is GRFS as a time to event endpoint from randomization. All randomized patients will be followed for one year; however, the primary endpoint will be analyzed as a time to event endpoint. The primary analysis will be done using the randomized population. An event for this time to event outcome is defined as grade III-IV acute GVHD, chronic GVHD requiring systemic immune suppression, disease relapse or progression, or death by any cause, whichever comes first. Time to event analyses were conducted. An unadjusted Kaplan-Meier analysis was done. Additionally, a multivariate Cox regression model adjusting for the following pre-specified covariates: age group (< 65 vs. 65+), disease risk index (low, intermediate, high/very high), planned RIC conditioning regimen (Fludarabine/Busulfan, Fludarabine/Melphalan, Other), donor type/HLA matching score (related 6/6, unrelated 7/8, unrelated 8/8), and planned use of post-transplant maintenance therapy (Yes vs. no).
Time Frame: 1 year post randomization
Population: Analysis Population includes all randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 214 | 217
percentage of participants | 52.3 [45.2 to 58.8] | 35.5 [29.1 to 42.0]
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the result of the Cox proportional hazards analysis. The null hypothesis is that there is no difference of GRFS hazard ratio between treatment groups after adjustment for age group, donor type and HLA Matching Score, disease risk index, Planned RIC Conditioning Regimen, and Planned post-transplant maintenance therapies; Test type: Superiority; p = 0.001, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05; Hazard Ratio (HR) = 0.641, 95% CI 2-sided [0.492 to 0.835]

2. Secondary Outcome: Percentage of Participants With Grades II-IV and III-IV Acute GVHD at Day 100 Post-transplant
Description: Acute GVHD was graded according to Mount Sinai aGVHD International Consortium (MAGIC) Criteria (Harris et al. 2016) with higher grade indicating worse outcomes. Grade I aGVHD is defined as Skin stage 1-2 and stage 0 for both GI and liver. Grade II is stage 3 skin, stage 1 GI, or stage 1 liver. Grade III is stage 2-3 GI or stage 2-3 liver. Grade IV is stage 4 skin or stage 4 liver. The cumulative incidence of acute GVHD grade II-IV and III-IV at Day 100 was estimated using the Aalen-Johansen estimator with 95% confidence intervals, treating death prior to aGVHD as a competing event. The cumulative incidences of Minnesota standard and high risk aGVHD at Day 100 were determined with 95% confidence intervals. Time to aGVHD is defined as time from transplant until onset of grades II-IV and III-IV aGVHD, respectively. A multivariate Cox regression model was used to compare the treatment groups, with adjustment for same baseline characteristics as for the primary endpoint.
Time Frame: Days 100 post-transplant
Population: Analysis Population includes transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
percentage of participants
  MAGIC aGVHD Grade II-IV | 53.8 [46.7 to 60.4] | 51.9 [44.9 to 58.4]
  MAGIC aGVHD Grade III-IV | 6.3 [3.5 to 10.2] | 14.7 [10.3 to 19.8]
  Standard risk aGVHD | 64.1 [57.1 to 70.3] | 64.3 [57.4 to 70.4]
  High risk aGVHD | 13.1 [8.9 to 18.1] | 18.5 [13.6 to 24.0]
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the unadjusted analysis. The null hypothesis is that there is no difference of grade II-IV acute GVHD post-transplantation between the treatment groups; Test type: Superiority; p = 0.995, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the unadjusted analysis. The null hypothesis is that there is no difference of grade III-IV acute GVHD post-transplantation between the treatment groups; Test type: Superiority; p = 0.001, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 3: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the result of the Cox proportional hazards analysis. The null hypothesis is that there is no difference of grade II-IV acute GVHD post-transplantation between the treatment groups using a Cox regression model for the cause-specific hazard of aGVHD; Test type: Superiority; p = 0.879, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05; Hazard Ratio (HR) = 0.980, 95% CI 2-sided [0.758 to 1.267]
Statistical Analysis 4: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the result of the Cox proportional hazards analysis. The null hypothesis is that there is no difference of grade III-IV aGVHD hazard ratio between treatment groups after adjustment for age group, donor type and HLA Matching Score, disease risk index, Planned RIC Conditioning Regimen, and Planned post-transplant maintenance therapies; Test type: Superiority; p = 0.001, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05; Hazard Ratio (HR) = 0.386, 95% CI 2-sided [0.215 to 0.691]

3. Secondary Outcome: Participants With Maximum Acute GVHD at One Year Post-transplant
Description: Acute GVHD were graded according to Mount Sinai Acute GVHD International Consortium (MAGIC) Criteria (Harris et al. Biology of Blood and Marrow Transplantation 2016; 22:4-10). The higher acute GVHD grade indicates worse outcomes. Grade 0 is no acute GVHD of any organ. Grade I acute GVHD is defined as Skin stage of 1-2 and stage 0 for both GI and liver organs. Grade II is stage 3 of skin, or stage 1 of GI, or stage 1 of liver. Grade III is stage 2-3 for GI, or stage 2-3 of liver. Grade IV is stage 4 of skin, or stage 4 of liver. Max acute GVHD by one-year post-transplant was computed.
Time Frame: One year post-transplant
Population: Analysis Population includes transplanted participants
Measure: Count of Participants; unit: Participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
Participants
  Grade 0 | 66 | 60
  Grade I | 27 | 32
  Grade II | 99 | 81
  Grade III | 11 | 25
  Grade IV | 5 | 14

4. Secondary Outcome: Participants With Maximum Stage of Skin, Lower GI, and Liver at Day 100 Post-transplant
Description: Organ stages were graded according to Mount Sinai Acute GVHD International Consortium (MAGIC) Criteria (Harris et al. 2016). Higher stage in any organ indicates worse outcomes. For skin, stage 0-no GVHD rash; 1-Maculopapular Rash <25% BSA; 2-Maculopapular Rash 25-50% BSA; 3-Maculopapular Rash >50% BSA; 4-Generalized Erythroderma Plus Bullous Formation and Desquamation >5% BSA. For Lower GI, 0-No Diarrhea or Diarrhea-Adult: <500 mL/day, <3 Episodes/day; Child: <10 mL/kg/day, <4 Episodes/day; 1-Diarrhea-Adult: 500-999 mL/day, 3-4 Episodes/day; Child: 10-19.9 mL/kg/day, 4-6 Episodes/day; 2-Diarrhea-Adult: 1000-1500 mL/day, 5-7 Episodes/day; Child: 20-30 mL/kg/day, 7-10 Episodes/day; 3-Diarrhea-Adult: >1500 mL/day, >7 Episodes/day; Child: >30 mL/kg/day, >10 Episodes/day; 4-Severe Abdominal Pain With or Without Ileus or Grossly Bloody Stool. For liver, 0-Bilirubin <2.0 mg/dL; 1-Bilirubin 2.0-3.0 mg/dL; 2-Bilirubin 3.1-6.0 mg/dL; 3-Bilirubin 6.1-15.0 mg/dL; 4-Bilirubin >15.0 mg/dL
Time Frame: Day 100 post-transplant
Population: Analysis Population includes transplanted participants
Measure: Count of Participants; unit: Participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
Participants
  Skin: 0 | 121 | 125
  Skin: 1 | 54 | 40
  Skin: 2 | 16 | 18
  Skin: 3 | 14 | 21
  Skin: 4 | 3 | 8
  Lower GI: 0 | 155 | 159
  Lower GI: 1 | 33 | 27
  Lower GI: 2 | 9 | 11
  Lower GI: 3 | 10 | 11
  Lower GI: 4 | 1 | 4
  Liver: 0 | 198 | 192
  Liver: 1 | 9 | 7
  Liver: 2 | 0 | 8
  Liver: 3 | 1 | 5
  Liver: 4 | 0 | 0

5. Secondary Outcome: Participants With Maximum Stage of Upper GI at Day 100 Post-transplant
Description: Organ stages were graded according to Mount Sinai Acute GVHD International Consortium (MAGIC) Criteria (Harris et al. 2016). Higher stage in any organ indicates worse outcomes. For upper GI, stage 0 is no or intermittent nausea, vomiting, or anorexia; stage 1 is persistent nausea, vomiting, or anorexia. The maximum stages of Upper GI at patient level were summarized at Day 100.
Time Frame: Day 100 post-transplant
Population: Analysis Population includes transplanted participants
Measure: Count of Participants; unit: Participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
Participants
  0 | 136 | 137
  1 | 72 | 75

6. Secondary Outcome: Percentage of Participants With Chronic GVHD Post-transplant
Description: Percentage of participants with chronic GVHD (cGVHD) at one-year will be estimated with 95% confidence intervals for each treatment group using the cumulative incidence estimate with the complementary log-log transformation, treating death prior to cGVHD as a competing event. Chronic GVHD is based on NIH Consensus Criteria (2014 NIH Consensus Criteria) and includes mild, moderate and severe chronic GVHD. Eight organs were scored on a 0-3 scale to reflect degree of cGVHD involvement. Liver and pulmonary function test results and use of systemic therapy for treatment of cGVHD were also recorded. Assessment of cGVHD occurred up to one-year post-transplant. This endpoint considers any cGVHD onset. A multivariate Cox regression model for the cause-specific hazard of cGVHD was used to compare the treatment groups, after adjustment for baseline characteristics as described for the primary endpoint.
Time Frame: 6, 12 months post-transplant
Population: Analysis Population includes transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
percentage of participants
  6 months post transplant | 11.3 [7.4 to 16.1] | 13.9 [9.6 to 19.0]
  12 months post transplant | 21.9 [16.4 to 27.9] | 35.1 [28.7 to 41.6]
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the unadjusted analysis. The null hypothesis is that there is no difference of chronic GVHD post-transplantation between the treatment groups; Test type: Superiority; p = 0.005, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the result of the Cox proportional hazards analysis. The null hypothesis is that there is no difference of the chronic GVHD hazard ratio between treatment groups after adjustment for age group, donor type and HLA Matching Score, disease risk index, Planned RIC Conditioning Regimen, and Planned post-transplant maintenance therapies; Test type: Superiority; p = 0.002, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05; Hazard Ratio (HR) = 0.556, 95% CI 2-sided [0.381 to 0.813]

7. Secondary Outcome: Number of Participants Experiencing Chronic GVHD With Maximum Severity at 12 Months Post-transplant
Description: Chronic GVHD data were collected directly from providers and chart review as defined by the NIH Consensus Conference Criteria. Eight organs were scored on a 0-3 scale to reflect degree of chronic GVHD involvement per the NIH global severity scores of mild, moderate and severe chronic GVHD. The maximum severity of chronic GVHD through 12 months post-transplant will be tabulated by treatment arm.
Time Frame: 12 months post-transplant
Population: Analysis Population includes transplanted participants
Measure: Count of Participants; unit: Participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
Participants
  None | 164 | 139
  Mild | 29 | 36
  Moderate | 11 | 24
  Severe | 3 | 11
  Unknown | 1 | 2

8. Secondary Outcome: Number of Participants With Immunosuppression-Free Survival (ISFS) at 1 Year Post-transplant
Description: Participants who are alive, relapse-free, and do not need ongoing immune suppression (IS) to control GVHD at one year post-transplant are considered successes for the endpoint immunosuppression-free survival (ISFS). Immune suppression is defined as any systemic agents used to control or suppress GVHD. Corticosteroid doses greater than 10 mg were considered active systemic immune suppression treatment. Participants who discontinued immune suppression within 15 days or less prior to the 1-year time point was considered to be on immune suppression for this endpoint.
Time Frame: 1 year post-transplant
Population: Analysis Population includes transplanted and evaluable participants for ISFS
Measure: Count of Participants; unit: Participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 198 | 204
Participants
  Immunosuppression-Free Survival | 99 | 81
  Death | 46 | 56
  Alive & Relapse | 21 | 22
  Alive, no relapse, and still on IS | 32 | 45

9. Secondary Outcome: Percentage of Participants With Immunosuppression-Free Survival (ISFS) at 1 Year Post-transplant
Description: Participants who are alive, relapse-free, and do not need ongoing immune suppression to control GVHD at one year post-transplant are considered successes for the endpoint immunosuppression-free survival (ISFS). Percentage of participants alive, relapse free, and off immune suppression at 1 year post-transplant were described for each treatment group, along with 95% Clopper-Pearson confidence intervals.
Time Frame: 1 year post-transplant
Population: Analysis Population includes transplanted and evaluable participants for ISFS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
percentage of participants | 50 [42.8 to 57.2] | 39.7 [32.9 to 42.8]
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; The null hypothesis is that there is no difference of Immunosuppression-Free Survival between the treatment groups; Test type: Superiority; p = 0.038, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05

10. Secondary Outcome: Percentage of Participants With Neutrophil Recovery Post-transplant
Description: Neutrophil recovery is defined as achieving an absolute neutrophil count (ANC) greater than or equal to 500/mm^3 for three consecutive measurements on three different days. The first of the three days will be designated the day of neutrophil recovery. The competing event is death without neutrophil recovery. For participants who never drop ANC below 500/mm^3, the date of neutrophil recovery will be Day +1 post-transplant. The cumulative incidence of neutrophil recovery by Day 28 and Day 100 was described for each treatment group with point estimates and 95% confidence intervals using the complementary log-log transformation and treating death as a competing event.
Time Frame: Days 28 and day 100 post-transplant
Population: Analysis Population includes transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
percentage of participants
  Day 28 post-transplant | 90.3 [85.3 to 93.6] | 93.4 [89.0 to 96.1]
  Day 100 post-transplant | 92.7 [88.1 to 95.6] | 97.2 [93.6 to 98.8]
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; The null hypothesis is that there is no difference of Neutrophil Recovery between the treatment groups; Test type: Superiority; p = 0.032, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05

11. Secondary Outcome: Percentage of Participants With Platelet Recovery Post-transplant
Description: Platelet recovery is defined by two different metrics: the first day of a sustained platelet count greater than or equal to 20,000/mm^3 or greater than or equal to 50,000/mm^3 with no platelet transfusions in the preceding seven days. The first day of sustained platelet count above these thresholds will be designated the day of platelet engraftment. For participants who never drop their platelet count below 20,000/mm^3 or 50,000/mm^3, the date of platelet recovery will be Day +1 post HCT. The competing event is death without platelet recovery. The cumulative incidence estimate of platelet recovery by Day 60 and Day 100 were described by treatment group with 95% confidence intervals (complementary log-log transformation), treating death as a competing event.
Time Frame: Day 60 and Day 100 post-transplant
Population: Analysis Population includes transplanted participants with platelet recovery data provided
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
percentage of participants
  Day 60 post-transplant of Platelet Recovery to >20k: number analyzed (Participants) | 207 | 208
  Day 60 post-transplant of Platelet Recovery to >20k | 88.3 [83.0 to 92.0] | 91.8 [87.1 to 94.8]
  Day 100 post-transplant of Platelet Recovery to >20k: number analyzed (Participants) | 207 | 208
  Day 100 post-transplant of Platelet Recovery to >20k | 90.3 [85.3 to 93.7] | 92.8 [88.2 to 95.6]
  Day 60 post-transplant of Platelet Recovery to >50k: number analyzed (Participants) | 206 | 208
  Day 60 post-transplant of Platelet Recovery to >50k | 77.6 [71.2 to 82.7] | 82.7 [76.8 to 87.2]
  Day 100 post-transplant of Platelet Recovery to >50k: number analyzed (Participants) | 206 | 208
  Day 100 post-transplant of Platelet Recovery to >50k | 79.5 [73.3 to 84.4] | 83.7 [77.9 to 88.1]
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; The null hypothesis is that there is no difference of Platelet Recovery greater than or equal to 20,000/mm^3 between the treatment groups; Test type: Superiority; p < 0.001, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; The null hypothesis is that there is no difference of Platelet Recovery greater than or equal to 50,000/mm^3 between the treatment groups; Test type: Superiority; p < 0.001, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05

12. Secondary Outcome: Percentage of Participants With Lymphocyte Recovery Post-transplant
Description: Lymphocyte recovery is defined as the first day of sustained absolute lymphocyte count greater than or equal to 1000/mm^3. The competing event is death without lymphocyte recovery. The cumulative incidence estimate of Lymphocyte recovery were described by treatment group with 95% confidence intervals (complementary log-log transformation), treating death as a competing event.
Time Frame: Day 60, Day 100, 6 Months, and 1 year post-transplant
Population: Analysis Population includes transplanted participants with lymphocyte recovery data provided.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
percentage of participants
  Day 60 post-transplant: number analyzed (Participants) | 208 | 210
  Day 60 post-transplant | 29.6 [23.5 to 35.9] | 48.2 [41.3 to 54.8]
  Day 100 post-transplant: number analyzed (Participants) | 208 | 210
  Day 100 post-transplant | 32.5 [26.2 to 39.0] | 52.5 [45.5 to 59.0]
  6 Months post-transplant: number analyzed (Participants) | 208 | 210
  6 Months post-transplant | 41.5 [34.7 to 48.2] | 58.3 [51.3 to 64.6]
  1 Year post-transplant: number analyzed (Participants) | 208 | 210
  1 Year post-transplant | 47.1 [40.1 to 53.8] | 63.2 [56.2 to 69.4]
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; The null hypothesis is that there is no difference of Lymphocyte Recovery between the treatment groups; Test type: Superiority; p < 0.001, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05

13. Secondary Outcome: Number of Participants With Each Level of Donor Cell Engraftment Post-transplant
Description: Donor cell engraftment were assessed with donor/recipient chimerism studies. Mixed chimerism is defined as the presence of donor cells, as a proportion of total cells to be less than 95% but at least 5% in the bone marrow or peripheral blood. Full donor chimerism is defined as greater than or equal to 95% of donor cells. Mixed and full chimerism will be evidence of donor cell engraftment. Donor cells of less than 5% will be considered as graft rejection. The number of participants with each level of chimerism described above is described as part of this outcome.
Time Frame: Day 28 and Day 100 post-transplant
Population: Analysis Population includes transplanted participants.
Measure: Count of Participants; unit: Participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
Participants
  Day 28 post-transplant: Full (>95% Donor Cells) | 126 | 129
  Day 28 post-transplant: Mixed (5-95% Donor Cells) | 39 | 45
  Day 28 post-transplant: Graft Rejection (<5% Donor Cells) | 4 | 4
  Day 28 post-transplant: Data missing | 39 | 34
  Day 100 post-transplant: Full (>95% Donor Cells) | 116 | 124
  Day 100 post-transplant: Mixed (5-95% Donor Cells) | 48 | 58
  Day 100 post-transplant: Graft Rejection (<5% Donor Cells) | 5 | 1
  Day 100 post-transplant: Data missing | 39 | 29
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; The null hypothesis is that there is no difference of Donor Cell Engraftment at Day 28 after transplantation between the treatment groups; Test type: Superiority; p = 0.919, Fisher Exact — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; The null hypothesis is that there is no difference of Donor Cell Engraftment at Day 100 after transplantation between the treatment groups; Test type: Superiority; p = 0.198, Fisher Exact — Statistical significance was determined using a pre-specified threshold of 0.05

14. Secondary Outcome: Summary Statistics for Donor Chimerism
Description: Donor cell engraftment were assessed with donor/recipient chimerism studies. Mixed chimerism is defined as the presence of donor cells, as a percentage of total cells to be less than 95% but at least 5% in the bone marrow or peripheral blood. Full donor chimerism is defined as greater than or equal to 95% of donor cells. Mixed and full chimerism will be evidence of donor cell engraftment. Donor cells of less than 5% will be considered as graft rejection. Donor chimerism at Day 28 and Day 100 after transplant in each of the randomized treatment arms will be described numerically as median and range for those evaluable.
Time Frame: Day 28 and Day 100 post-transplant
Population: Analysis Population includes transplanted participants who submitted post-transplant assessments.
Measure: Median (Full Range); unit: percentage of donor cells
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
percentage of donor cells
  Day 28 post-transplant: number analyzed (Participants) | 169 | 178
  Day 28 post-transplant | 100 [0 to 100] | 100 [0 to 100]
  Day 100 post-transplant: number analyzed (Participants) | 169 | 183
  Day 100 post-transplant | 99 [0 to 100] | 99 [4 to 100]
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; The null hypothesis is that there is no difference of quantitative donor chimerism at Day 28 after transplantation between the treatment groups; Test type: Superiority; p = 0.670, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; The null hypothesis is that there is no difference of quantitative donor chimerism at Day 100 after transplantation between the treatment groups; Test type: Superiority; p = 0.607, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

15. Secondary Outcome: Percentage of Participants With Disease Relapse at 1 Year Post-transplant
Description: Disease relapse/progression is defined as being alive and free of relapse/progression of the primary disease. The time from transplant until relapse/progression of the primary disease, or cumulative incidence, was estimated at one-year post-transplant along with 95% CIs computed using the complementary log-log transformation, treating death prior to disease relapse as a competing event. A multivariate Cox regression model for the cause-specific hazard of relapse or progression will be used to compare the treatment groups, after adjustment for baseline characteristics as described for the primary endpoint.
Time Frame: 1 year post-transplant
Population: Analysis Population includes transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
percentage of participants | 20.8 [15.5 to 26.7] | 20.2 [15.0 to 25.9]
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the unadjusted analysis. The null hypothesis is that there is no difference of Disease Relapse between the treatment groups; Test type: Superiority; p = 0.906, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the result of the Cox proportional hazards analysis. The null hypothesis is that there is no difference of Disease Relapse hazard ratio between treatment groups after adjustment for age group, donor type and HLA Matching Score, disease risk index, Planned RIC Conditioning Regimen, and Planned post-transplant maintenance therapies; Test type: Superiority; p = 0.947, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05; Hazard Ratio (HR) = 0.985, 95% CI 2-sided [0.641 to 1.515]

16. Secondary Outcome: Percentage of Participants With Treatment-related Mortality (TRM) Post-transplant
Description: An event for this endpoint TRM is death without evidence of disease progression or recurrence. Disease progression or recurrence will be considered a competing event. The time from transplant until TRM, or cumulative incidence, estimated at specific time points along with 95% CIs computed using the complementary log-log transformation, treating relapse/progression of the primary disease as a competing risk. A multivariate Cox regression model for the cause-specific hazard of TRM was used to compare the treatment groups, after adjustment for baseline characteristics as described for the primary endpoint.
Time Frame: Days 100, 180 and 1 year post-transplant
Population: Analysis Population includes transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
percentage of participants
  Day 100 post-transplant | 6.8 [3.9 to 10.8] | 7.6 [4.5 to 11.7]
  Day 180 post-transplant | 8.8 [5.4 to 13.2] | 13.3 [9.1 to 18.3]
  12 Months post-transplant | 12.3 [8.2 to 17.2] | 17.2 [12.4 to 22.6]
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the unadjusted analysis. The null hypothesis is that there is no difference of Treatment-related Mortality between the treatment groups; Test type: Superiority; p = 0.167, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the result of the Cox proportional hazards analysis. The null hypothesis is that there is no difference of Treatment-related Mortality hazard ratio between treatment groups after adjustment for age group, donor type and HLA Matching Score, disease risk index, Planned RIC Conditioning Regimen, and Planned post-transplant maintenance therapies; Test type: Superiority; p = 0.133, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05; Hazard Ratio (HR) = 0.675, 95% CI 2-sided [0.404 to 1.127]

17. Secondary Outcome: Number of Participants Reporting Grade 3-5 Toxicities by 1 Year Post-transplant
Description: All Grade 3-5 toxicities will be tabulated by grade for each randomized treatment arm, by type of toxicity as well as the peak grade overall. Toxicities were evaluated using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Time Frame: 1 year post-transplant
Population: Analysis Population includes transplanted participants
Measure: Count of Participants; unit: Participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
Participants
  Grades 3-5 General Disorders | 51 | 48
  Grades 3-5 Immune System Disorders | 5 | 6
  Grades 3-5 GI Disorders | 57 | 77
  Grades 3-5 Renal Disorders | 33 | 30
  Grades 3-5 Hemorrhagic Disorders | 12 | 11
  Grades 3-5 Cardiac Disorders | 71 | 72
  Grades 3-5 Nervous System Disorders | 12 | 20
  Grades 3-5 Blood and Lymphatic Disorders | 3 | 3
  Grades 3-5 Vascular Disorders | 6 | 12
  Grades 3-5 Musculoskeletal and Connective Tissue Disorders | 17 | 12
  Grades 3-5 Respiratory, Thoracic and Mediastinal Disorders | 41 | 42
  Grades 3-5 Metabolism and Nutrition Disorders | 24 | 33
  Grades 3-5 Hepatic Disorders | 24 | 44
  Received Dialysis | 11 | 8
  Hepatitis | 6 | 4
  Liver failure | 2 | 4
  Abnormal liver function | 14 | 15
  Overall Grade 3 | 141 | 146
  Overall Grade 4 | 23 | 27
  Overall Grade 5 | 12 | 11
  Maximum Toxicity Grade 3 | 113 | 116
  Maximum Toxicity Grade 4 | 17 | 22
  Maximum Toxicity Grade 5 | 12 | 11

18. Secondary Outcome: Frequencies of Infections Categorized by Infection Type
Description: All Grade 2 and 3 infections were reported according to the BMT CTN Technical Manual of Procedures (MOP) up to 1 year post-transplant. The frequency of Grade 2-3 infections and the number of participants experiencing infections occurring within 1 year post-transplant, are tabulated by treatment arm, organism, time period of infection onset, and severity, with Grade defined per the BMT CTN Technical MOP.
Time Frame: 1 year post-transplant
Population: Analysis Population includes transplanted participants
Measure: Number; unit: infections
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
infections
  Bacterial | 128 | 118
  Viral | 70 | 61
  Fungal | 18 | 14
  Protozoal/Parasite | 0 | 0
  Other | 34 | 46

19. Secondary Outcome: Number of Participants With Grade 2 and 3 Infections
Description: as for outcome 18
Time Frame: 1 year post-transplant
Population: Analysis Population includes transplanted participants
Measure: Count of Participants; unit: Participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
Participants
  Patients with Infections | 109 | 100
  Patients with 1 Infection | 46 | 46
  Patients with 2 Infections | 32 | 24
  Patients with 3 Infections | 14 | 10
  Patients with 4 Infections | 8 | 7
  Patients with 5 Infections | 4 | 5
  Patients with >= 6 Infections | 5 | 8
  Maximum Severity of None | 99 | 112
  Maximum Severity of Grade 1 | 21 | 19
  Maximum Severity of Grade 2 | 57 | 36
  Maximum Severity of Grade 3 | 25 | 28
  CMV Reactivation by Day 100 | 15 | 16
  Non-Microbial Infections | 9 | 10

20. Secondary Outcome: Percentage of Participants With Grade 2 and 3 Infections
Description: Grade 2 and 3 infections, as defined by the BMT CTN Technical Manual of Procedures (MOP), are reported on the study. The cumulative incidence of infections post transplantation, treating death as a competing risk, were compared between the treatment groups using the Gray's test.
Time Frame: 6 months and 1 year post-transplant
Population: Analysis Population includes transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
percentage of participants
  6 months post-transplant | 36.4 [29.8 to 43.0] | 24.1 [18.6 to 30.1]
  1 year post-transplant | 40.0 [33.2 to 46.7] | 30.4 [24.3 to 36.7]
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; The null hypothesis is that there is no difference of Grade 2 and 3 infections between the treatment groups; Test type: Superiority; p = 0.018, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05

21. Secondary Outcome: Percentage of Participants With CMV at Day 100 Post-transplant
Description: The cumulative incidence of initiation of systemic treatment for CMV was compared between the treatment groups using the Gray's test, with death treated as a competing risk. Estimates of the cumulative incidence of CMV reactivation are provided at Day 100 post-transplant.
Time Frame: Day 100 post-transplant
Population: Analysis Population includes transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
percentage of participants | 7.3 [4.3 to 11.4] | 7.1 [4.1 to 11.1]
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; The null hypothesis is that there is no difference of CMV between the treatment groups; Test type: Superiority; p = 0. 825, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05

22. Secondary Outcome: Percentage of Participants With Disease-Free Survival (DFS) at 1 Year Post-transplant
Description: DFS is defined as being alive and free of relapse/progression of the primary disease. The time from transplant until death or relapse/progression (DFS failure) was described for each treatment arm using the Kaplan-Meier estimator, with numbers of subjects at risk at specific time points presented for each treatment group. A multivariate Cox regression model for the hazard of death will be used to compare the treatment groups, after adjustment for baseline characteristics as described for the primary endpoint.
Time Frame: 1 year post-transplant
Population: Analysis Population includes transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
percentage of participants | 67.0 [60.0 to 73.0] | 62.6 [55.7 to 68.8]
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the unadjusted analysis. The null hypothesis is that there is no difference of Disease-Free Survival between the treatment groups; Test type: Superiority; p = 0.351, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the result of the Cox proportional hazards analysis. The null hypothesis is that there is no difference of Disease-Free Survival hazard ratio between treatment groups after adjustment for age group, donor type and HLA Matching Score, disease risk index, Planned RIC Conditioning Regimen, and Planned post-transplant maintenance therapies; Test type: Superiority; p = 0.320, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05; Hazard Ratio (HR) = 0.847, 95% CI 2-sided [0.610 to 1.176]

23. Secondary Outcome: Percentage of Participants With Overall Survival (OS) at 1 Year Post-transplant
Description: The event for this endpoint OS is death from any cause post-transplant. Time to overall survival is defined as the time interval between date of transplant and date of death from any cause. Surviving participants will be censored at last follow-up or 1 year post-transplant, whichever comes first. The time from transplant until death from any cause was described graphically for each treatment arm using the Kaplan-Meier estimator, with numbers of subjects at risk at specific time points presented for each treatment group. A multivariate Cox regression model for the hazard of death will be used to compare the treatment groups, after adjustment for baseline characteristics as described for the primary endpoint.
Time Frame: 1 year post-transplant
Population: Analysis Population includes transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
percentage of participants | 76.8 [70.3 to 82.0] | 72.6 [66.0 to 78.2]
Statistical Analysis 1: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the unadjusted analysis. The null hypothesis is that there is no difference of Overall Survival between the treatment groups; Test type: Superiority; p = 0.335, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: PTCY/Tacrolimus/MMF vs Tacrolimus/Methotrexate; This is the result of the Cox proportional hazards analysis. The null hypothesis is that there is no difference of the Overall Survival hazard ratio between treatment groups after adjustment for age group, donor type and HLA Matching Score, disease risk index, Planned RIC Conditioning Regimen, and Planned post-transplant maintenance therapies; Test type: Superiority; p = 0.252, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05; Hazard Ratio (HR) = 0.797, 95% CI 2-sided [0.541 to 1.175]

24. Secondary Outcome: Percentage of Participants With Lymphoproliferative Disease (PTLD) at 1 Year Post-Transplant
Description: The cumulative incidence of lymphoproliferative disease at 1-year post-transplant is described with 95% confidence intervals for each treatment group using the Aalen-Johansen estimator, treating death as a competing event.
Time Frame: 1 year Post-Transplant
Population: Analysis Population includes transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
Number analyzed (Participants) | 208 | 212
percentage of participants | 0.5 [0 to 2.6] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Deaths were assessed for all randomized participants. Adverse Events were assessed only for participants who underwent transplant throughout the study, an average of 1 year. More deaths are reported in the AE module than that in the secondary outcome section because deaths reported in the AE module were counted starting at randomization and throughout the study, whereas deaths reported in survival analysis were counted starting at transplant and throughout one-year post-transplant.
Description: AE reporting was conducted according to the BMT CTN's Manual of Operating Procedures. Unexpected, serious AEs (SAEs) were reported through an expedited AE reporting system. Expected AEs were reported using National Cancer Institute (NCI)'s Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 at regular intervals. Any expected life-threatening SAE not collected as toxicities were reported through the expedited AE reporting system.
Arm/Group | PTCY/Tacrolimus/MMF | Tacrolimus/Methotrexate
All-Cause Mortality (participants affected / at risk) | 58/214 | 70/217
Serious Adverse Events (participants affected / at risk) | 7/208 | 14/212
Other Adverse Events (participants affected / at risk) | 142/208 | 149/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTCY/Tacrolimus/MMF (N=208) | Tacrolimus/Methotrexate (N=212)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Homicide (Social circumstances) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTCY/Tacrolimus/MMF (N=208) | Tacrolimus/Methotrexate (N=212)
Grades 3-5 General Disorders (General disorders) | 51 (68) | 48 (61)
Grades 3-5 Immune System Disorders (Immune system disorders) | 5 (5) | 6 (6)
Grades 3-5 GI Disorders (Gastrointestinal disorders) | 57 (73) | 77 (116)
Grades 3-5 Renal Disorders (Renal and urinary disorders) | 33 (46) | 30 (42)
Grades 3-5 Hemorrhagic Disorders (Vascular disorders) | 12 (13) | 11 (11)
Grades 3-5 Cardiac Disorders (Cardiac disorders) | 71 (117) | 72 (125)
Grades 3-5 Nervous System Disorders (Nervous system disorders) | 12 (13) | 20 (25)
Grades 3-5 Blood and Lymphatic Disorders (Blood and lymphatic system disorders) | 3 (4) | 3 (4)
Grades 3-5 Vascular Disorders (Vascular disorders) | 6 (7) | 12 (13)
Grades 3-5 Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 17 (18) | 12 (15)
Grades 3-5 Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 41 (58) | 42 (52)
Grades 3-5 Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 24 (31) | 33 (51)
Grades 3-5 Hepatic Disorders (Hepatobiliary disorders) | 24 (30) | 44 (54)
Received Dialysis (Renal and urinary disorders) | 11 (17) | 8 (11)
Hepatitis (Hepatobiliary disorders) | 6 (8) | 4 (9)
Liver failure (Hepatobiliary disorders) | 2 (2) | 4 (4)
Abnormal liver function (Hepatobiliary disorders) | 14 (19) | 15 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT03959241/Prot_001.pdf
  • Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT03959241/SAP_002.pdf
  • Informed Consent Form (2021-01-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT03959241/ICF_003.pdf